CLINICAL TRIAL: NCT01098812
Title: Clinical Evaluation of the TECNIS® Toric 1-Piece Intraocular Lens
Brief Title: Clinical Evaluation of a 1-Piece Intraocular Lens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIOL-103-TCNS
Record Dates: First submitted 2010-03-31; First posted 2010-04-05 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract
Keywords: Cataract, Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control IOL (Active Comparator): Approved Intraocular control lens
  Interventions: Device: Tecnis ZCB00 IOL (control)
- Toric IOL (Experimental): Investigational Toric IOL
  Interventions: Device: Toric Intraocular lens
- Higher Cylinder Toric IOL (Experimental): Investigational Toric IOLs with higher cylinder powers.
  Interventions: Device: Toric Intraocular lens

INTERVENTIONS:
Device: Tecnis ZCB00 IOL (control) — Tecnis 1-piece acrylic IOL
  Arms: Control IOL
Device: Toric Intraocular lens — Toric acrylic intraocular lens with various cylinder powers
  Arms: Higher Cylinder Toric IOL; Toric IOL

SUMMARY:
The aims of this study are to:

* Demonstrate a reduction in postoperative cylinder compared to results from the control lens
* Demonstrate better uncorrected distance visual acuity compared to the control lens

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Cataract for which phacoemulsification extraction and posterior chamber IOL implantation has been planned for both eyes
* Preoperative best corrected distance visual acuity (BCDVA)of 20/40 or worse (Snellen), with or without glare, for each eye
* BCDVA projected to be better than 20/30 following cataract removal and IOL implantation for each eye
* Preoperative keratometric cylinder of 0.75 diopters to 3.62 diopters for each eye (with exception of second eyes with 0.0-0.75 diopters planned to receive non-toric IOL)
* Clear intraocular media other than cataract in both eyes
* Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits
* Signed informed consent and HIPAA authorization

Exclusion Criteria:

* Requiring IOLs outside spherical power range of +15.0 to +28.0 diopters
* Dilated pupil size less than 5.5 mm or the presence of any pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)in either eye
* Previous corneal or intraocular surgery in either eye
* Irregular corneal astigmatism in either eye
* Corneal pathology/abnormality potentially affecting topography in either eye
* Corneal abnormalities such as stromal, epithelial or endothelial dystrophies in either eye
* Inability to achieve keratometric stability in either eye for contact lens wearers
* Subjects with diagnosed degenerative visual disorders in either eye(eg., macular degeneration or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma, or posterior capsule defects
* An eccentric anterior capsulorhexis, zonular damage/rupture or capsular tear/rupture during the cataract extraction procedure
* Use of systemic or ocular medications that may affect vision
* Prior, current, or anticipated use during the course of the nine month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo)likely to affect dilation or iris structure
* Poorly-controlled diabetes
* Acute, chronic, or uncontrolled systemic disease or illness that would, in the opinion of the investigator, increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, etc.)
* Uncontrolled ocular hypertension or glaucomatous changes in the retina or visual field in either eye
* Known ocular disease or pathology that may affect visual acuity or that may require surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation or participation during 30 days prior to preoperative visit in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, O.D., Study Director — Abbott Medical Optics

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from normal cataract populations at 14 investigative sites.
Pre-assignment Details: Subjects with low cylinder were enrolled in a randomized group and received either the control lens or the investigational Toric IOL. Subjects with higher cylinder were enrolled in the high cylinder group and received a higher cylinder investigational Toric IOL.
Groups:
- ZCB00: Approved Intraocular control lens
Period: Overall Study
Arm/Group | ZCB00 | Toric IOL | Higher Cylinder Toric IOL
Started | 95 | 102 | 72
Completed | 93 | 101 | 71
Not Completed | 2 | 1 | 1
Not completed — Death | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZCB00 | Toric IOL | Higher Cylinder Toric IOL | Total
Number analyzed (Participants) | 95 | 102 | 72 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (9) | 70 (8) | 69 (9) | 70 (9)
Age, Customized [Number; unit: participants]
  <60 years | 5 | 10 | 7 | 22
  60 through 69 years | 36 | 39 | 33 | 108
  70 through 79 years | 36 | 41 | 25 | 102
  >=80 years | 18 | 12 | 7 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 40 | 150
  Male | 40 | 47 | 32 | 119
Region of Enrollment [Number; unit: participants]
  United States | 87 | 94 | 66 | 247
  Canada | 8 | 8 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Reduction in Cylinder
Description: Reduction in cylinder postoperatively vs. preoperatively (baseline) as measured by keratometry and manifest refraction. Mean percent reduction in cylinder = (postoperative refractive cylinder minus preoperative keratometric cylinder)/(target refractive cylinder minus preoperative keratometric cylinder). Reduction in cylinder was assessed in the first eye (per participant) for contribution to the mean.
Time Frame: 6 months after second eye implant compared to baseline
Population: Subjects at the final visit with preoperative keratometric cylinder, intended/target cylinder and postoperative refractive cylinder.
Measure: Mean (Standard Deviation); unit: percentage of reduction in cylinder
Arm/Group | Control IOL | Toric IOL | Higher Cylinder Toric IOL
Number analyzed (Participants) | 91 | 101 | 70
percentage of reduction in cylinder | 32 (79) | 75 (72) | 76. (33)
Statistical Analysis 1: Comparison: Control IOL vs Toric IOL; Toric IOL results for mean percent reduction in cyl compared to control results at 6 months. Null hypothesis = mean reduction for toric eyes is <= to that of control eyes; alternate hypothesis = mean reduction for toric eyes is > the control. There is 80% power to detect >=31% difference in mean percent reduction in cylinder (postoperative refractive cylinder minus preoperative keratometric cylinder)/(target refractive cylinder minus preoperative keratometric cylinder) between IOL groups; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — Primary study endpoint; therefore, no adjustment for multiple comparisons. The planned alpha level for testing was 0.025; Mean Difference (Final Values) = 43, 90% CI 1-sided [lower limit 25], Standard Deviation 75

2. Secondary Outcome: Uncorrected Distance Visual Acuity (UCDVA)
Description: Postoperative uncorrected distance visual acuity as measured by LogMAR acuity. For comparison: LogMAR value of 0.0 = Snellen 20/20; LogMar 0.10 = Snellen 20/25; LogMAR 0.20 = Snellen 20/32; LogMAR 0.30 = Snellen 20/40. Uncorrected distance visual acuity as measured by LogMAR acuity was assessed in the first eye (per participant) for contribution to the mean.
Time Frame: 6 months after second eye implant
Population: Available subjects at the final visit with measured uncorrected distance visual acuity.
Measure: Mean (Standard Deviation); unit: LogMAR acuity values
Arm/Group | Control IOL | Toric IOL | Higher Cylinder Toric IOL
Number analyzed (Participants) | 93 | 101 | 71
LogMAR acuity values | 0.16 (0.16) | 0.10 (0.14) | 0.11 (0.12)
Statistical Analysis 1: Comparison: Control IOL vs Toric IOL; Used LogMAR values for visual acuity; The null hypothesis is that the mean UCDVA for toric eyes is worse than or equal to that for control eyes; the alternate hypothesis is that the mean UCDVA for toric eyes is better than that for control eyes. There is 80% power to detect >=0.06 LogMAR difference in mean UCDVA between IOL groups; Test type: Superiority or Other; p = 0.0009, t-test, 1 sided — P-value compared to alpha level adjusted for multiplicity of 0.0125; Mean Difference (Final Values) = -0.07, 90% CI 1-sided [upper limit -0.03], Standard Deviation 0.15

ADVERSE EVENTS:
Groups:
- All Toric IOLs: Investigational Toric IOLs including high cylinder powers
Arm/Group | ZCB00 | All Toric IOLs
Serious Adverse Events (participants affected / at risk) | 0/95 | 6/174
Other Adverse Events (participants affected / at risk) | 0/95 | 0/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZCB00 (N=95) | All Toric IOLs (N=174)
Lens Repositioning Procedure (Eye disorders) | 0 (0) | 4 (4)
Retinal Repair (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results may be published by PI upon written approval by sponsor (AMO). Any proposed submission for publication or presentation of study data must be provided to AMO 90 days prior to submission for review, comment and approval. Sponsor may delay or withhold submission as necessary (ongoing study activities, patents pending, etc.).